CLINICAL TRIAL: NCT01473433
Title: Randomized Trial to Evaluate the Safety and Efficacy of a New Surgical Approach to Cardiac Regeneration: Pericardic Adipose Pedicle Transposition Over the Myocardial Infarct (adiFLAP Trial)
Brief Title: Pericardic Adipose Pedicle Transposition Over the Myocardial Infarct (adiFLAP Trial)
Acronym: adiFLAP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Antoni Bayés Genís, Chief of the Cardiology Service, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ICREC-2011-02
Record Dates: First submitted 2011-11-14; First posted 2011-11-17 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Myocardial Infarction
Keywords: Regenerative medicine; Myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control (Other): Patients in which the non-revascularizable area will be left untouched and the revascularizable area will be treated normally.
  Interventions: Other: Control
- adiFLAP (Experimental): Patients in which the non-revascularizable area will be covered by the adiFLAP and the revascularizable area will be treated with the normal procedure.
  Interventions: Procedure: Pericardial adipose pedicle (adiFLAP) transposition.

INTERVENTIONS:
Procedure: Pericardial adipose pedicle (adiFLAP) transposition. — Patients with a established transmural necrosis, candidates for revascularization of other myocardial areas, will be enrolled. The non-revascularizable area will be covered by the adiFLAP and the revascularizable area will be treated with the normal procedure. A non-revascularizable area will be considered whenever a transmural necrosis is detected by means of gadolinium contrast using MRI.
  Arms: adiFLAP
Other: Control — Patients with a established transmural necrosis, candidates for revascularization of other myocardial areas, will be enrolled. The non-revascularizable area will be left untouched and the revascularizable area will be treated normally (by-pass).
  Arms: Control

SUMMARY:
The purpose of this trial is to evaluate safety and efficacy of a pericardial adipose pedicle transposition (adiFLAP) for the improvement of cardiac function in patients with a chronic myocardial infarct. Preclinical studies in the porcine model of myocardial infarction have shown that AdiFLAP reduces infarct area.

DETAILED DESCRIPTION:
This novel intervention consists of the pericardial isolation of adipose tissue maintaining its vascularization to create an adipose flap (adiFLAP) and its transposition fully covering infarcted myocardium.

ELIGIBILITY:
Inclusion Criteria:

* Established transmural myocardial infarction non candidate to revascularization (>3 months-old)
* Candidate to coronary by-pass for other territories different from the previous transmural infarct.
* > 18 years of age, male or female, capable of giving an informed consent.

Exclusion Criteria:

* Severe co-morbidity associated with a reduction in life expectancy of less than 1 year.
* Severe valvular disease candidate for surgical restoration.
* Candidate to ventricular remodeling.
* Contraindication for NMR (creatinin clearance <30 ml/min/1.73m2, metallic implants, claustrophobia).
* Severe renal or hepatic failure.
* Abnormal laboratory tests (no explanation at the time of inclusion).
* Previous cardiac intervention.
* High surgical risk (Euroscore 2).
* Pregnant or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Appearance of adverse effects derived from the procedure (7 days after the surgical procedure and 1 year follow-up). | 12 months

SECONDARY OUTCOMES:
Improvement of cardiac function as changes in clinical variables, cardiac magnetic resonance imaging and echocardiography, and biochemical variables (NTproBNP and high sensitivity troponin T). | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Germans Trias Research Institute; Germans Trias University Hospital, Badalona, Barcelona, Spain

REFERENCES:
- [Background] Galvez-Monton C, Prat-Vidal C, Roura S, Farre J, Soler-Botija C, Llucia-Valldeperas A, Diaz-Guemes I, Sanchez-Margallo FM, Aris A, Bayes-Genis A. Transposition of a pericardial-derived vascular adipose flap for myocardial salvage after infarct. Cardiovasc Res. 2011 Sep 1;91(4):659-67. doi: 10.1093/cvr/cvr136. Epub 2011 May 16. PMID 21576133
- [Background] Galvez-Monton C, Prat-Vidal C, Roura S, Soler-Botija C, Llucia-Valldeperas A, Diaz-Guemes I, Sanchez-Margallo FM, Bayes-Genis A. Post-infarction scar coverage using a pericardial-derived vascular adipose flap. Pre-clinical results. Int J Cardiol. 2013 Jun 20;166(2):469-74. doi: 10.1016/j.ijcard.2011.11.019. Epub 2011 Dec 2. PMID 22137092
- [Derived] Bayes-Genis A, Gastelurrutia P, Camara ML, Teis A, Lupon J, Llibre C, Zamora E, Alomar X, Ruyra X, Roura S, Revilla A, San Roman JA, Galvez-Monton C. First-in-man Safety and Efficacy of the Adipose Graft Transposition Procedure (AGTP) in Patients With a Myocardial Scar. EBioMedicine. 2016 May;7:248-54. doi: 10.1016/j.ebiom.2016.03.027. Epub 2016 Apr 10. PMID 27322478